CLINICAL TRIAL: NCT01159938
Title: The Effect of Postprandial Hyperglycemia on the Arterial Stiffness in Patients With Type 2 Diabetes
Brief Title: A Study of Postprandial Hyperglycemia in Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 13087; F3Z-EW-IOPT (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-06-17; First posted 2010-07-12 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- T2DM, albuminuria but normal kidney function (Experimental)
  Interventions: Drug: Lispro
- Healthy participants (No Intervention)
- T2DM, normal urinary albumin excretion rate (UAER) (Experimental)
  Interventions: Drug: Lispro

INTERVENTIONS:
Drug: Lispro — Dosage based on participants with type 2 diabetes mellitus (T2DM) normal morning insulin dose and energy content of participant's normal breakfast. Subcutaneous injection given on one occasion. Administered once on low post prandial day.
  Other Names: Humalog; LY275585
  Arms: T2DM, albuminuria but normal kidney function; T2DM, normal urinary albumin excretion rate (UAER)

SUMMARY:
This Study is looking at whether high blood glucose levels after a meal affect arterial stiffness more or less than low blood glucose levels, and whether certain cardiovascular markers influence the outcome of this.

ELIGIBILITY:
Inclusion Criteria:

* Are diagnosed with T2DM (according to the American Diabetes Association classification [American Diabetes Association 2006]) and on insulin therapy for at least 6 months.
* Have not smoked in the last 12 hours prior to the study visit.
* Have albuminuria but normal kidney function or normal UAER [UAER < 20 micrograms per minute (mcg/min) or < 30 milligrams/24 hours (mg/24h), respectively]. Participants with or without albuminuria but normal kidney function will be matched for age and body mass index (BMI).
* Participants have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests and examinations required by the protocol.
* Each participant must understand the nature of the study and must sign an informed consent document (ICD).

Healthy participants are eligible to be included in the study only if they meet all of the following criteria:

* Healthy participants 45 to 70 years of age, matched for age and BMI, who have not smoked in the last 12 hours prior to the study.
* Normal glucose tolerance and normal UAER (UAER between < 20 μg/min in the overnight urine collection or < 30 mg/24h in the 24-h urine collection).
* Healthy participants have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests and examinations required by the protocol.
* Each healthy participant must understand the nature of the study and must sign an ICD.

Exclusion Criteria:

Participants/healthy participants will be excluded from the study if they meet any of the following criteria:

* Have had a cardiovascular event [stroke, myocardial infarction (MI), coronary artery procedure (by-pass surgery or angioplasty), limb amputation due to ischemia, peripheral vascular disease] or coronary heart disease confirmed by exercise test or scintigraphy.
* Have arrhythmias.
* Have an acute infection.
* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational drug or device or off-label use of a drug or device (other than the study drug/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Are unwilling or unable to comply with the use of a data collection device to directly record data from the participant.

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM to 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Helsinki, Finland

REFERENCES:
- [Derived] Gordin D, Saraheimo M, Tuomikangas J, Soro-Paavonen A, Forsblom C, Paavonen K, Steckel-Hamann B, Harjutsalo V, Nicolaou L, Pavo I, Koivisto V, Groop PH. Insulin exposure mitigates the increase of arterial stiffness in patients with type 2 diabetes and albuminuria: an exploratory analysis. Acta Diabetol. 2019 Nov;56(11):1169-1175. doi: 10.1007/s00592-019-01351-4. Epub 2019 May 22. PMID 31119456
- [Derived] Gordin D, Saraheimo M, Tuomikangas J, Soro-Paavonen A, Forsblom C, Paavonen K, Steckel-Hamann B, Vandenhende F, Nicolaou L, Pavo I, Koivisto V, Groop PH. Influence of Postprandial Hyperglycemic Conditions on Arterial Stiffness in Patients With Type 2 Diabetes. J Clin Endocrinol Metab. 2016 Mar;101(3):1134-43. doi: 10.1210/jc.2015-3635. Epub 2016 Jan 5. PMID 26731258
- [Derived] Muka T, de Jonge EA, Kiefte-de Jong JC, Uitterlinden AG, Hofman A, Dehghan A, Zillikens MC, Franco OH, Rivadeneira F. The Influence of Serum Uric Acid on Bone Mineral Density, Hip Geometry, and Fracture Risk: The Rotterdam Study. J Clin Endocrinol Metab. 2016 Mar;101(3):1113-22. doi: 10.1210/jc.2015-2446. Epub 2015 Dec 18. PMID 26684274

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with type 2 diabetes mellitus (T2DM) were randomized to either a high to low blood glucose sequence or a low to high blood glucose sequence dependent upon whether they received insulin lispro or not in the first study period. Participants were stratified into treatment arms based on their urinary albumin excretion rate (UAER).
Groups:
- Healthy Participants: Healthy participants with normal glucose tolerance and normal UAER did not receive an insulin lispro subcutaneous injection but participated in study assessments. Normal glucose tolerance according to World Health Organization (WHO) criteria was defined as fasting glucose <6.1 millimoles/liter (mmol/L) and 2-hour glucose <7.8 mmol/L. Normal UAER was defined as <20 micrograms per minute (mcg/min) of albumin in the overnight urine collection or <30 milligrams per 24 hours (mg/24h) of albumin in the 24-hour urine collection.
- T2DM With Albuminuria, High to Low: T2DM participants with abnormal UAER [albuminuria (defined as urinary albumin)] but normal kidney function who did not receive an insulin lispro subcutaneous injection in the first study period and who received an insulin lispro subcutaneous injection prior to a standard breakfast in the second study period. The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
- T2DM With Albuminuria, Low to High: T2DM participants with abnormal UAER (albuminuria) but normal kidney function who received an insulin lispro subcutaneous injection prior to a standard breakfast in the first study period and who did not receive an insulin lispro subcutaneous injection in the second study period. The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
- T2DM With Normal UAER, High to Low: T2DM participants with normal UAER who did not receive an insulin lispro subcutaneous injection in the first study period and who received an insulin lispro subcutaneous injection prior to a standard breakfast in the second study period. The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
- T2DM With Normal UAER, Low to High: T2DM participants with normal UAER who received an insulin lispro subcutaneous injection prior to a standard breakfast in the first study period and who did not receive an insulin lispro subcutaneous injection in the second study period. The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
Period: First Study Period
Arm/Group | Healthy Participants | T2DM With Albuminuria, High to Low | T2DM With Albuminuria, Low to High | T2DM With Normal UAER, High to Low | T2DM With Normal UAER, Low to High
Started | 26 | 11 | 11 | 12 | 12
Received at Least 1 Dose of Study Drug | 0 | 11 | 11 | 12 | 12
Safety and Efficacy Analysis Population | 25 (One healthy participant completed study but was excluded from analyses (major protocol violation).) | 11 | 11 (Microalbuminuria relaxed with protocol amendment. T2DM albuminuria participant included in analyses.) | 12 | 12
Completed | 26 | 11 | 10 | 12 | 12
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation (Microalbuminuria) | 0 | 0 | 1 | 0 | 0
Period: Second Study Period
Arm/Group | Healthy Participants | T2DM With Albuminuria, High to Low | T2DM With Albuminuria, Low to High | T2DM With Normal UAER, High to Low | T2DM With Normal UAER, Low to High
Started | 0 | 11 | 10 | 12 | 12
Completed | 0 | 11 | 10 | 12 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants, with the exception of 1 healthy participant who completed the study but was later excluded from analyses due to major protocol violation.
Groups:
- Healthy Participants: Healthy participants with normal glucose tolerance and normal urinary albumin excretion rate (UAER) did not receive an insulin lispro subcutaneous injection but participated in study assessments. Normal glucose tolerance according to World Health Organization (WHO) criteria was defined as fasting glucose <6.1 millimoles/liter (mmol/L) and 2-hour glucose <7.8 mmol/L. Normal UAER was defined as <20 micrograms per minute (mcg/min) of albumin in the overnight urine collection or <30 milligrams per 24 hours (mg/24h) of albumin in the 24-hour urine collection.
- T2DM With Albuminuria: T2DM participants with abnormal UAER [albuminuria (defined as urinary albumin)] but normal kidney function who received an insulin lispro subcutaneous injection prior to a standard breakfast in the first study period and who did not receive an insulin lispro subcutaneous injection prior to standard breakfast in the second study period (low to high sequence) or participants who did not receive an insulin lispro subcutaneous injection prior to a standard breakfast in the first study period and who received an insulin lispro subcutaneous injection prior to a standard breakfast in the second study period (high to low sequence). The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
- T2DM With Normal UAER: T2DM participants with normal UAER who received an insulin lispro subcutaneous injection prior to a standard breakfast in the first study period and who did not receive an insulin lispro subcutaneous injection prior to a standard breakfast in the second study period (low to high sequence) or participants who did not receive an insulin lispro subcutaneous injection prior to a standard breakfast in the first study period and who received an insulin lispro subcutaneous injection prior to a standard breakfast in the second study period (high to low sequence). The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | T2DM With Albuminuria | T2DM With Normal UAER | Total
Number analyzed (Participants) | 25 | 22 | 24 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (6.6) | 61.2 (4.9) | 63.7 (5.2) | 61.2 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 25 | 22 | 24 | 71
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25 | 22 | 24 | 71
Region of Enrollment [Number; unit: participants]
  Finland | 25 | 22 | 24 | 71

OUTCOME MEASURES:

1. Primary Outcome: Postprandial Pulse Wave Velocity (PWV) in Type 2 Diabetes Mellitus (T2DM) Participants at 30 Minutes (Mins) Pre-Breakfast
Description: The PWV measured arterial stiffness in the aortic and brachial arteries of T2DM participants. The Least Square (LS) mean was estimated from a mixed-effect analysis of covariance (ANCOVA) model that was adjusted for age, body mass index (BMI), visit, group, condition, group by condition, and random participant.
Time Frame: 30 mins (pre-breakfast)
Population: Randomized T2DM participants who were scheduled to receive study drug and had a baseline PWV measurement at the specified time point and no major protocol deviation.
Measure: Least Squares Mean (95% Confidence Interval); unit: meters per second (m/s)
Groups:
- T2DM Overall (High Postprandial Glucose): T2DM participants with normal urinary albumin excretion rate (UAER) and T2DM participants with abnormal UAER [albuminuria (defined as urinary albumin)] but normal kidney function who did not receive an insulin lispro subcutaneous injection prior to a standard breakfast either in the first or second study period (high postprandial glucose day). Normal UAER was defined as <20 micrograms per minute (mcg/min) of albumin in the overnight urine collection or <30 milligrams per 24 hours (mg/24h) of albumin in the 24-hour urine collection.
- T2DM Overall (Low Postprandial Glucose): T2DM participants with normal UAER and T2DM participants with abnormal UAER (albuminuria) but normal kidney function who were scheduled to receive an insulin lispro subcutaneous injection prior to a standard breakfast in the first or second study period (low postprandial glucose day). The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
- T2DM With Albuminuria (High Postprandial Glucose): T2DM participants with abnormal UAER (albuminuria) but normal kidney function who did not receive an insulin lispro subcutaneous injection prior to a standard breakfast either in the first or second study period (high postprandial glucose day).
- T2DM With Albuminuria (Low Postprandial Glucose): T2DM participants with abnormal UAER (albuminuria) but normal kidney function who were scheduled to receive an insulin lispro subcutaneous injection prior to a standard breakfast in the first or second study period (low postprandial glucose day). The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
- T2DM With Normal UAER (High Postprandial Glucose): T2DM participants with normal UAER who did not receive an insulin lispro subcutaneous injection prior to a standard breakfast either in the first or second study period (high postprandial glucose day).
- T2DM With Normal UAER (Low Postprandial Glucose): T2DM participants with normal UAER who were scheduled to receive an insulin lispro subcutaneous injection prior to a standard breakfast in the first or second study period (low postprandial glucose day). The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
Arm/Group | T2DM Overall (High Postprandial Glucose) | T2DM Overall (Low Postprandial Glucose) | T2DM With Albuminuria (High Postprandial Glucose) | T2DM With Albuminuria (Low Postprandial Glucose) | T2DM With Normal UAER (High Postprandial Glucose) | T2DM With Normal UAER (Low Postprandial Glucose)
Number analyzed (Participants) | 45 | 45 | 21 | 22 | 24 | 23
meters per second (m/s)
  Aortic PWV (n=44, 44, 21, 22, 23, 22) | 10.99 [9.98 to 11.99] | 10.73 [9.72 to 11.73] | 11.56 [10.08 to 13.04] | 11.31 [9.86 to 12.75] | 10.41 [9.01 to 11.81] | 10.15 [8.71 to 11.59]
  Brachial PWV (n=45, 45, 21, 22, 24, 23) | 7.49 [7.02 to 7.96] | 7.84 [7.37 to 8.30] | 7.79 [7.10 to 8.48] | 7.99 [7.32 to 8.67] | 7.19 [6.54 to 7.84] | 7.68 [7.02 to 8.34]
Statistical Analysis 1: Comparison: T2DM Overall (High Postprandial Glucose) vs T2DM Overall (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.617, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 30-min pre-breakfast in aortic arteries. Significance was assessed at the 2-sided 5% level; LS mean difference = 0.26, 95% CI 2-sided [-0.78 to 1.30]
Statistical Analysis 2: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.732, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.25, 95% CI 2-sided [-1.23 to 1.73]
Statistical Analysis 3: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.715, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.27, 95% CI 2-sided [-1.20 to 1.73]
Statistical Analysis 4: Comparison: T2DM Overall (High Postprandial Glucose) vs T2DM Overall (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.177, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 30-min pre-breakfast in brachial arteries. Significance was assessed at 2-sided 5% level; LS Mean Difference = -0.35, 95% CI 2-sided [-0.85 to 0.16]
Statistical Analysis 5: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.579, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 30-min pre-breakfast in brachial arteries. Significance was assessed at the 2-sided 5% level; LS Mean Difference = -0.20, 95% CI 2-sided [-0.94 to 0.53]
Statistical Analysis 6: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.167, ANCOVA — [p-value comment as in outcome 1, analysis 4]; LS Mean Difference = -0.49, 95% CI 2-sided [-1.19 to 0.21]

2. Primary Outcome: Postprandial Pulse Wave Velocity (PWV) in Type 2 Diabetes Mellitus (T2DM) Participants at 60 Minutes (Mins) Post-Breakfast
Description: as for outcome 1
Time Frame: 60 mins (post-breakfast)
Population: Randomized T2DM participants who received study drug and had a post-baseline PWV measurement at the specified time point and no major protocol deviation.
Measure: Least Squares Mean (95% Confidence Interval); unit: meters per second (m/sec)
Groups:
- T2DM Overall (Low Postprandial Glucose): T2DM participants with normal UAER and T2DM participants with abnormal UAER (albuminuria) but normal kidney function who received an insulin lispro subcutaneous injection prior to a standard breakfast in the first or second study period (low postprandial glucose day). The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
- T2DM With Albuminuria (Low Postprandial Glucose): T2DM participants with abnormal UAER (albuminuria) but normal kidney function who received an insulin lispro subcutaneous injection prior to a standard breakfast in the first or second study period (low postprandial glucose day). The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
- T2DM With Normal UAER (Low Postprandial Glucose): T2DM participants with normal UAER who received an insulin lispro subcutaneous injection prior to a standard breakfast in the first or second study period (low postprandial glucose day). The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
Arm/Group | T2DM Overall (High Postprandial Glucose) | T2DM Overall (Low Postprandial Glucose) | T2DM With Albuminuria (High Postprandial Glucose) | T2DM With Albuminuria (Low Postprandial Glucose) | T2DM With Normal UAER (High Postprandial Glucose) | T2DM With Normal UAER (Low Postprandial Glucose)
Number analyzed (Participants) | 45 | 45 | 21 | 22 | 24 | 23
meters per second (m/sec)
  Aortic PWV (n= 44, 45, 21, 22, 23, 23) | 10.19 [9.38 to 11.00] | 10.38 [9.57 to 11.18] | 10.26 [9.06 to 11.45] | 10.22 [9.06 to 11.38] | 10.12 [8.98 to 11.25] | 10.53 [9.39 to 11.67]
  Brachial PWV (n=45, 45, 21, 22, 24, 23) | 7.71 [7.27 to 8.16] | 7.80 [7.36 to 8.25] | 8.03 [7.37 to 8.69] | 8.00 [7.36 to 8.65] | 7.39 [6.78 to 8.01] | 7.61 [6.98 to 8.23]
Statistical Analysis 1: Comparison: T2DM Overall (High Postprandial Glucose) vs T2DM Overall (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.676, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 60-min post-breakfast in aortic arteries. Significance was assessed at the 2-sided 5% level; LS Mean Difference = -0.19, 95% CI 2-sided [-1.10 to 0.72]
Statistical Analysis 2: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.957, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 0.03, 95% CI 2-sided [-1.27 to 1.34]
Statistical Analysis 3: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.513, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = -0.41, 95% CI 2-sided [-1.68 to 0.85]
Statistical Analysis 4: Comparison: T2DM Overall (High Postprandial Glucose) vs T2DM Overall (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.623, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 60-min post-breakfast in brachial arteries. Significance was assessed at the 2-sided 5% level; LS Mean Difference = -0.09, 95% CI 2-sided [-0.47 to 0.28]
Statistical Analysis 5: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.916, ANCOVA — [p-value comment as in outcome 2, analysis 4]; LS Mean Difference = 0.03, 95% CI 2-sided [-0.51 to 0.57]
Statistical Analysis 6: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.413, ANCOVA — [p-value comment as in outcome 2, analysis 4]; LS Mean Difference = -0.21, 95% CI 2-sided [-0.73 to 0.31]

3. Primary Outcome: Postprandial Pulse Wave Velocity (PWV) in Type 2 Diabetes Mellitus (T2DM) Participants at 120 Minutes (Mins) Post-Breakfast
Description: as for outcome 1
Time Frame: 120 mins (post-breakfast)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: meters per second (m/sec)
Arm/Group | T2DM Overall (High Postprandial Glucose) | T2DM Overall (Low Postprandial Glucose) | T2DM With Albuminuria (High Postprandial Glucose) | T2DM With Albuminuria (Low Postprandial Glucose) | T2DM With Normal UAER (High Postprandial Glucose) | T2DM With Normal UAER (Low Postprandial Glucose)
Number analyzed (Participants) | 45 | 45 | 21 | 22 | 24 | 23
meters per second (m/sec)
  Aortic PWV (n=45, 44, 21, 22, 24, 22) | 10.96 [9.83 to 12.10] | 10.76 [9.62 to 11.91] | 11.18 [9.50 to 12.87] | 10.61 [8.96 to 12.26] | 10.74 [9.17 to 12.32] | 10.92 [9.28 to 12.56]
  Brachial PWV (n=45, 45, 21, 22, 24, 23) | 7.66 [7.19 to 8.14] | 7.86 [7.38 to 8.34] | 7.84 [7.13 to 8.54] | 8.03 [7.33 to 8.72] | 7.49 [6.83 to 8.16] | 7.70 [7.02 to 8.37]
Statistical Analysis 1: Comparison: T2DM Overall (High Postprandial Glucose) vs T2DM Overall (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.724, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 120-min post-breakfast in aortic arteries. Significance was assessed at the 2-sided 5% level; LS Mean Difference = 0.20, 95% CI 2-sided [-0.94 to 1.34]
Statistical Analysis 2: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.479, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 120-min post-breakfast in aortic arteries. Significance was assessed at 2-sided 5% level; LS Mean Difference = 0.57, 95% CI 2-sided [-1.05 to 2.20]
Statistical Analysis 3: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.825, ANCOVA — [p-value comment as in outcome 3, analysis 2]; LS Mean Difference = -0.18, 95% CI 2-sided [-1.76 to 1.41]
Statistical Analysis 4: Comparison: T2DM Overall (High Postprandial Glucose) vs T2DM Overall (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.378, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 120-min post-breakfast in brachial arteries. Significance was assessed at the 2-sided 5% level; LS Mean Difference = -0.20, 95% CI 2-sided [-0.65 to 0.25]
Statistical Analysis 5: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.553, ANCOVA — The p-value is for the LS mean difference (high minus low postprandial glucose) in PWV at 120 mins post-breakfast in brachial arteries. Significance was assessed at the 2-sided 5% level; LS Mean Difference = -0.19, 95% CI 2-sided [-0.84 to 0.46]
Statistical Analysis 6: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.512, ANCOVA — [p-value comment as in outcome 3, analysis 4]; LS Mean Difference = -0.20, 95% CI 2-sided [-0.83 to 0.42]

4. Primary Outcome: Postprandial Pulse Wave Velocity (PWV) in Type 2 Diabetes Mellitus (T2DM) Participants at 180 Minutes (Mins) Post-Breakfast
Description: as for outcome 1
Time Frame: 180 mins (post-breakfast)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: meters per second (m/sec)
Arm/Group | T2DM Overall (High Postprandial Glucose) | T2DM Overall (Low Postprandial Glucose) | T2DM With Albuminuria (High Postprandial Glucose) | T2DM With Albuminuria (Low Postprandial Glucose) | T2DM With Normal UAER (High Postprandial Glucose) | T2DM With Normal UAER (Low Postprandial Glucose)
Number analyzed (Participants) | 45 | 45 | 21 | 22 | 24 | 23
meters per second (m/sec)
  Aortic PWV (n= 45, 45, 21, 22, 24, 23) | 10.99 [9.99 to 12.00] | 11.28 [10.28 to 12.29] | 11.04 [9.55 to 12.52] | 11.47 [10.01 to 12.94] | 10.95 [9.55 to 12.35] | 11.09 [9.67 to 12.51]
  Brachial PWV (n= 45, 45, 21, 22, 24, 23) | 7.75 [7.29 to 8.22] | 7.91 [7.45 to 8.38] | 7.75 [7.06 to 8.44] | 8.32 [7.65 to 9.00] | 7.76 [7.11 to 8.41] | 7.50 [6.84 to 8.16]
Statistical Analysis 1: Comparison: T2DM Overall (High Postprandial Glucose) vs T2DM Overall (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.466, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 180-min post-breakfast in aortic arteries. Significance was assessed at the 2-sided 5% level; LS Mean Difference = -0.29, 95% CI 2-sided [-1.09 to 0.51]
Statistical Analysis 2: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.449, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -0.44, 95% CI 2-sided [-1.60 to 0.72]
Statistical Analysis 3: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.792, ANCOVA — [p-value comment as in outcome 4, analysis 1]; LS Mean Difference = -0.15, 95% CI 2-sided [-1.25 to 0.96]
Statistical Analysis 4: Comparison: T2DM Overall (High Postprandial Glucose) vs T2DM Overall (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.493, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 180-min post-breakfast in brachial arteries. Significance was assessed at the 2-sided 5% level; LS Mean Difference = -0.16, 95% CI 2-sided [-0.63 to 0.31]
Statistical Analysis 5: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.091, ANCOVA — [p-value comment as in outcome 4, analysis 4]; LS Mean Difference = -0.58, 95% CI 2-sided [-1.25 to 0.10]
Statistical Analysis 6: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.425, ANCOVA — [p-value comment as in outcome 4, analysis 4]; LS Mean Difference = 0.26, 95% CI 2-sided [-0.39 to 0.90]

5. Primary Outcome: Postprandial Pulse Wave Velocity (PWV) in Type 2 Diabetes Mellitus (T2DM) Participants at 240 Minutes (Mins) Post-Breakfast
Description: as for outcome 1
Time Frame: 240 mins (post-breakfast)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: meters per second (m/sec)
Arm/Group | T2DM Overall (High Postprandial Glucose) | T2DM Overall (Low Postprandial Glucose) | T2DM With Albuminuria (High Postprandial Glucose) | T2DM With Albuminuria (Low Postprandial Glucose) | T2DM With Normal UAER (High Postprandial Glucose) | T2DM With Normal UAER (Low Postprandial Glucose)
Number analyzed (Participants) | 45 | 45 | 21 | 22 | 24 | 23
meters per second (m/sec)
  Aortic PWV (n= 45, 45, 21, 22, 24, 23) | 11.09 [10.09 to 12.09] | 11.57 [10.57 to 12.57] | 10.99 [9.50 to 12.47] | 11.16 [9.70 to 12.62] | 11.19 [9.79 to 12.58] | 11.98 [10.56 to 13.39]
  Brachial PWV (n= 45, 45, 21, 22, 24, 23) | 7.76 [7.28 to 8.24] | 8.16 [7.68 to 8.64] | 7.99 [7.28 to 8.70] | 8.42 [7.72 to 9.11] | 7.53 [6.86 to 8.20] | 7.90 [7.22 to 8.58]
Statistical Analysis 1: Comparison: T2DM Overall (High Postprandial Glucose) vs T2DM Overall (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.275, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 240-min post-breakfast in aortic arteries. Significance was assessed at the 2-sided 5% level; LS Mean Difference = -0.48, 95% CI 2-sided [-1.36 to 0.40]
Statistical Analysis 2: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.784, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -0.17, 95% CI [-1.44 to 1.10]
Statistical Analysis 3: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.197, ANCOVA — [p-value comment as in outcome 5, analysis 1]; LS Mean Difference = -0.79, 95% CI 2-sided [-2.01 to 0.43]
Statistical Analysis 4: Comparison: T2DM Overall (High Postprandial Glucose) vs T2DM Overall (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.122, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in PWV at 240-min post-breakfast in brachial arteries. Significance was assessed at the 2-sided 5% level; LS Mean Difference = -0.40, 95% CI 2-sided [-0.90 to 0.11]
Statistical Analysis 5: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.246, ANCOVA — [p-value comment as in outcome 5, analysis 4]; LS Mean Difference = -0.43, 95% CI 2-sided [-1.16 to 0.31]
Statistical Analysis 6: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.298, ANCOVA — [p-value comment as in outcome 5, analysis 4]; LS Mean Difference = -0.37, 95% CI 2-sided [-1.06 to 0.33]

6. Secondary Outcome: Change in Pulse Wave Amplitude (PWA)
Description: The PWA measured systemic arterial stiffness (augmentation index). PWA was reported as a percentage of systolic peak and calculated as the difference between second and first systolic peak in an ascending aortic pulse pressure waveform divided by the first systolic peak then multiplied by 100. The change in PWA from baseline [30-minute (min) pre-breakfast] is reported.
Time Frame: 30 mins (pre-breakfast), 60, 120, 180 and 240 mins (post-breakfast)
Population: Enrolled healthy and randomized type 2 diabetes mellitus (T2DM) participants with a baseline and a post-baseline PWA measurement at specified time point and no major protocol deviation.
Measure: Mean (Standard Deviation); unit: percentage of systolic peak
Groups:
- T2DM With Albuminuria (High Postprandial Glucose): T2DM participants with abnormal UAER [albuminuria (defined as urinary albumin)] but normal kidney function who did not receive an insulin lispro subcutaneous injection prior to a standard breakfast either in the first or second study period (high postprandial glucose day).
Arm/Group | Healthy Participants | T2DM With Albuminuria (High Postprandial Glucose) | T2DM With Albuminuria (Low Postprandial Glucose) | T2DM With Normal UAER (High Postprandial Glucose) | T2DM With Normal UAER (Low Postprandial Glucose)
Number analyzed (Participants) | 25 | 21 | 22 | 24 | 24
percentage of systolic peak
  60-Min Post-Breakfast | -4.4 (5.19) | -4.1 (5.75) [16.53 to 22.65] | -0.6 (4.88) [17.78 to 23.82] | -2.3 (3.91) [15.13 to 20.92] | -2.5 (7.00) [15.50 to 21.29]
  120-Min Post-Breakfast | -2.9 (4.33) | -3.7 (5.09) [16.75 to 22.60] | -1.7 (6.81) [16.94 to 22.71] | -2.9 (4.45) [14.52 to 20.05] | -2.3 (6.80) [15.72 to 21.25]
  180-Min Post-Breakfast | -1.9 (6.41) | -2.3 (5.81) [18.13 to 24.24] | -0.5 (5.85) [18.11 to 24.13] | 1.0 (5.50) [18.17 to 23.94] | -1.1 (7.28) [16.74 to 22.52]
  240-Min Post-Breakfast | 2.1 (15.21) | -2.2 (5.31) [18.66 to 24.25] | 0.6 (4.73) [19.31 to 24.82] | -0.7 (4.95) [16.93 to 22.22] | -0.6 (6.34) [17.63 to 22.92]
Statistical Analysis 1: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.024, ANCOVA — P-value is for the Least Square (LS) mean difference (high minus low postprandial glucose) in change in PWA at 60-min post-breakfast. Significance was assessed at the 2-sided 5% level; LS mean was adjusted for age, body mass index (BMI), visit, group, condition, group by condition, and random participant; LS Mean Difference = -3.49, 95% CI 2-sided [-6.50 to -0.48]
Statistical Analysis 2: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.859, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in change in PWA at 60-min post-breakfast. Significance was assessed at the 2-sided 5% level; The LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = 0.25, 95% CI 2-sided [-2.59 to 3.09]
Statistical Analysis 3: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.155, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in change in PWA at 120-min post-breakfast. Significance was assessed at the 2-sided 5% level; LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = -2.19, 95% CI 2-sided [-5.25 to 0.87]
Statistical Analysis 4: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.685, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in change in PWA at 120-min post-breakfast. Significance was assessed at 2-sided 5% level; LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = -0.58, 95% CI 2-sided [-3.46 to 2.30]
Statistical Analysis 5: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.292, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in change in PWA at 180-min post-breakfast. Significance was assessed at the 2-sided 5% level; LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = -1.84, 95% CI 2-sided [-5.33 to 1.64]
Statistical Analysis 6: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.216, ANCOVA — [p-value comment as in outcome 6, analysis 5]; LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = 2.04, 95% CI 2-sided [-1.25 to 5.33]
Statistical Analysis 7: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.065, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in change in PWA at 240-min post-breakfast. Significance was assessed at the 2-sided 5% level; LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = -2.87, 95% CI 2-sided [-5.92 to 0.18]
Statistical Analysis 8: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.954, ANCOVA — [p-value comment as in outcome 6, analysis 7]; LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = -0.08, 95% CI 2-sided [-2.96 to 2.80]

7. Secondary Outcome: Change in Peripheral Artery Tonometry (PAT)
Description: The PAT device is a pneumatic plethysmograph that applies uniform pressure to the surface of each finger tip and measures digital pulse amplitude. The PAT was reported as a percentage of pulse amplitude and expressed as the ratio of post deflation to baseline pulse amplitude in hyperemic finger divided by the same ratio in the contralateral finger that served as a control. The change in PAT from baseline [30-minute (min) pre-breakfast] is reported.
Time Frame: 30 mins (pre-breakfast), 120 and 240 mins (post-breakfast)
Population: Enrolled healthy and randomized T2DM participants who had a baseline and a post-baseline PAT measurement at specified time point and no major protocol deviation.
Measure: Mean (Standard Deviation); unit: percentage of pulse amplitude
Arm/Group | Healthy Participants | T2DM With Albuminuria (High Postprandial Glucose) | T2DM With Albuminuria (Low Postprandial Glucose) | T2DM With Normal UAER (High Postprandial Glucose) | T2DM With Normal UAER (Low Postprandial Glucose)
Number analyzed (Participants) | 24 | 21 | 22 | 23 | 23
percentage of pulse amplitude
  120-Min Post-Breakfast (n= 23, 20, 22, 23, 23) | 0.03 (0.582) | 0.09 (0.490) [1.85 to 2.31] | 0.11 (0.445) [1.80 to 2.25] | 0.36 (0.543) [1.82 to 2.25] | -0.05 (0.597) [1.79 to 2.23]
  240-Min Post-Breakfast (n= 24, 21, 22, 23, 21) | 0.15 (0.634) | 0.23 (0.532) [1.91 to 2.42] | 0.32 (0.585) [1.99 to 2.49] | 0.36 (0.444) [1.80 to 2.28] | 0.24 (0.559) [2.04 to 2.55]
Statistical Analysis 1: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.905, ANCOVA — P-value is for Least Square (LS) mean difference (high minus low postprandial glucose) in change in PAT at 120-min post-breakfast. Significance was assessed at the 2-sided 5% level; LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = -0.02, 95% CI 2-sided [-0.31 to 0.27]
Statistical Analysis 2: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.004, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in change in PAT at 120-min post-breakfast. Significance was assessed at the 2-sided 5% level; LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = 0.42, 95% CI 2-sided [0.14 to 0.69]
Statistical Analysis 3: Comparison: T2DM With Albuminuria (High Postprandial Glucose) vs T2DM With Albuminuria (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.584, ANCOVA — P-value is for LS mean difference (high minus low postprandial glucose) in change in PAT at 240-min post-breakfast. Significance was assessed at the 2-sided 5% level; LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = -0.09, 95% CI 2-sided [-0.41 to 0.23]
Statistical Analysis 4: Comparison: T2DM With Normal UAER (High Postprandial Glucose) vs T2DM With Normal UAER (Low Postprandial Glucose); Test type: Superiority or Other; p = 0.436, ANCOVA — [p-value comment as in outcome 7, analysis 3]; LS mean was adjusted for age, BMI, visit, group, condition, group by condition, and random participant; LS Mean Difference = 0.13, 95% CI 2-sided [-0.19 to 0.44]

8. Secondary Outcome: Change in QT Interval on Electrocardiogram (ECG)
Description: QT interval is a measure of time from the beginning of the QRS complex to the end of the T wave on an ECG during which contraction of the ventricles occurs. Changes in QT interval from baseline [30-minute (min) pre-breakfast] are reported.
Time Frame: 30 mins (pre-breakfast), 60, 120, 180 and 240 mins (post-breakfast)
Population: Enrolled healthy and randomized type 2 diabetes mellitus (T2DM) participants who had a baseline and a post-baseline QT interval measurement at specified time point and no major protocol deviation.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Healthy Participants | T2DM With Albuminuria (High Postprandial Glucose) | T2DM With Albuminuria (Low Postprandial Glucose) | T2DM With Normal UAER (High Postprandial Glucose) | T2DM With Normal UAER (Low Postprandial Glucose)
Number analyzed (Participants) | 25 | 21 | 21 | 24 | 24
milliseconds (msec)
  60-Min Post-Breakfast (n=25, 20, 21, 24, 24) | 12.1 (11.71) | 23.8 (81.00) | 6.5 (9.12) | 11.0 (10.47) | 11.3 (14.73)
  120-Min Post-Breakfast (n=25, 21, 21, 24, 24) | -0.4 (12.29) | 18.0 (75.72) | -0.8 (5.74) | 1.4 (9.84) | 2.8 (10.89)
  180-Min Post-Breakfast (n=25, 21, 21, 23 ,24) | 8.3 (10.06) | 19.1 (77.11) | 5.8 (7.45) | 2.5 (9.80) | 4.5 (10.24)
  240-Min Post-Breakfast (n=25, 21, 21, 24, 24) | 10.4 (13.05) | 18.5 (75.04) | 7.2 (7.63) | 5.0 (9.67) | 5.6 (11.87)

9. Secondary Outcome: Change in Blood Glucose (BG)
Description: Changes in BG from the baseline [30-minute (min) pre-breakfast] are reported.
Time Frame: 30 mins (pre-breakfast), 50, 110 ,170, and 230 mins (post-breakfast)
Population: Enrolled healthy and randomized type 2 diabetes mellitus (T2DM) participants who had a baseline and a post-baseline blood glucose measurement at specified time point and no major protocol deviation.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Groups:
- Healthy Participants: Healthy participants with normal glucose tolerance and normal urinary albumin excretion rate (UAER) did not receive an insulin lispro subcutaneous injection but participated in study assessments. Normal glucose tolerance according to World Health Organization (WHO) criteria was defined as fasting glucose <6.1 millimoles/liter (mmol/L) and 2-hour glucose <7.8 mmol/L. Normal UAER was defined as <20 micrograms per minute (mcg/min) of albumin in the overnight urine collection or <30 milligrams albumin per 24 hours (mg/24h) of albumin in the 24-hour urine collection.
Arm/Group | Healthy Participants | T2DM With Albuminuria (High Postprandial Glucose) | T2DM With Albuminuria (Low Postprandial Glucose) | T2DM With Normal UAER (High Postprandial Glucose) | T2DM With Normal UAER (Low Postprandial Glucose)
Number analyzed (Participants) | 25 | 21 | 22 | 24 | 24
millimoles per liter (mmol/L)
  50-Min Post-Breakfast (n=24, 21, 22, 24, 24) | 0.07 (1.191) | 4.98 (1.546) | 3.39 (1.510) | 5.59 (2.338) | 3.23 (2.257)
  110-Min Post-Breakfast (n= 25, 21, 22, 24, 24) | -0.15 (0.729) | 4.73 (1.716) | 2.52 (1.723) | 5.58 (2.918) | 2.59 (2.561)
  170-Min Post-Breakfast (n= 25, 21, 22, 24, 24) | -0.36 (0.656) | 3.14 (2.013) | 0.29 (1.691) | 3.65 (3.071) | 1.26 (2.637)
  230-Min Post-Breakfast (n= 25, 21, 22, 24, 24) | -0.54 (0.412) | 1.78 (2.182) | -0.92 (1.788) | 1.79 (2.529) | -0.13 (2.124)

10. Secondary Outcome: Change in Postprandial Pulse Wave Velocity (PWV)
Description: The PWV measured arterial stiffness in the aortic and brachial arteries of healthy participants and T2DM participants. Changes in PWV from baseline [30-minute (min) pre-breakfast] are reported.
Time Frame: 30 mins (pre-breakfast), 60, 120, 180 and 240 mins (post-breakfast)
Population: Enrolled healthy and randomized type 2 diabetes mellitus (T2DM) participants who had a baseline and post-baseline PWV measurement at specified time point and no major protocol deviation.
Measure: Mean (Standard Deviation); unit: meters per second (m/sec)
Arm/Group | Healthy Participants | T2DM With Albuminuria (High Postprandial Glucose) | T2DM With Albuminuria (Low Postprandial Glucose) | T2DM With Normal UAER (High Postprandial Glucose) | T2DM With Normal UAER (Low Postprandial Glucose)
Number analyzed (Participants) | 24 | 21 | 22 | 24 | 23
meters per second (m/sec)
  60-Min Post-Breakfast (Aortic;n=22,21,22,23,22) | -0.26 (1.410) | -0.74 (3.244) | -0.91 (4.888) | -0.52 (2.031) | 0.22 (3.431)
  120-Min Post-Breakfast (Aortic;n=22,21,22,23,22) | 0.25 (1.400) | 0.04 (4.702) | -0.58 (3.392) | 0.09 (2.771) | 0.75 (3.124)
  180-Min Post-Breakfast (Aortic;n=23,21,22,23,22) | -0.00 (1.429) | -0.32 (3.326) | 0.22 (2.983) | 0.48 (2.514) | 0.94 (3.488)
  240-Min Post-Breakfast (Aortic;n=23,21,22,23,22) | 0.99 (1.372) | -0.09 (3.128) | 0.00 (3.972) | 0.61 (3.032) | 1.65 (3.730)
  60-Min Post-Breakfast (Brachial;n=23,21,22,24,23) | -0.13 (1.294) | 0.23 (1.399) | 0.03 (1.243) | 0.19 (1.495) | -0.06 (1.629)
  120-Min Post-Breakfast (Brachial;n=22,21,22,24,23) | 0.23 (1.176) | 0.09 (0.935) | 0.09 (1.352) | 0.25 (1.475) | -0.04 (1.567)
  180-Min Post-Breakfast (Brachial;n=24,21,22,24,23) | -0.37 (1.518) | -0.06 (1.394) | 0.35 (1.723) | 0.55 (1.694) | -0.23 (1.761)
  240-Min Post-Breakfast (Brachial;n=23,21,22,24,23) | -0.10 (1.475) | 0.17 (1.177) | 0.41 (1.402) | 0.35 (1.415) | 0.23 (1.682)

ADVERSE EVENTS:
Groups:
- T2DM With Albuminuria: T2DM participants with abnormal UAER [albuminuria(defined as urinary albumin)] but normal kidney function who received an insulin lispro subcutaneous injection prior to a standard breakfast in the first study period and who did not receive an insulin lispro subcutaneous injection prior to a standard breakfast in the second study period (low to high sequence) or participants who did not receive an insulin lispro subcutaneous injection prior to a standard breakfast in the first study period and who received an insulin lispro subcutaneous injection prior to a standard breakfast in the second study period (high to low sequence). The dosage of insulin lispro was adjusted as needed based on the energy content of the participant's normal breakfast and standard basal insulin dose.
Arm/Group | Healthy Participants | T2DM With Albuminuria | T2DM With Normal UAER
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/22 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days